CLINICAL TRIAL: NCT06066983
Title: Treating Anxiety in Young Children With Autism
Brief Title: DINO RCT - Treating Anxiety in Children With Autism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Responsible Party: Principal Investigator, Amy Keefer, Principal Investigator, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00343724; CDMRP - AR220066 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2023-09-28; First posted 2023-10-04 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-03

CONDITIONS: Autism Spectrum Disorder; Anxiety Disorders
MeSH Terms: conditions — Autism Spectrum Disorder; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Parent-child dyads will receive DINOSAUR, a group-based cognitive-behavioral therapy (CBT) intervention, adapted for young children and delivered via telehealth. This 14 week intervention teaches parents and children strategies to reduce anxiety and intolerance of uncertainty, an underlying construct of anxiety.
  Interventions: Behavioral: DINOSAUR
- Active Control (Active Comparator): Parents in the active control condition will participate in three psychoeducational groups focused on presenting information regarding anxiety prevalence, differentiating anxiety from autism, and anxiety triggers. These groups will be delivered via telehealth across a 14-week period.
  Interventions: Other: Psychoeducation

INTERVENTIONS:
Behavioral: DINOSAUR — This intervention aims to treat intolerance of uncertainty and anxiety in young autistic children.
  Arms: Treatment
Other: Psychoeducation — This intervention provides psychoeducation regarding anxiety and autism.
  Arms: Active Control

SUMMARY:
Anxiety is prevalent in young children, under 7 years of age, with autism. Yet, few studies have examined anxiety interventions for this age range, and only one anxiety treatment study has included young children with cognitive and language delays. Anxiety treatment models utilizing cognitive-behavioral therapy (CBT), adapted for children with autism, are empirically supported in school-age autistic children. Further, preliminary evidence suggests CBT approaches may reduce intolerance of uncertainty (IU), a mechanistic construct that may contribute to the maintenance of anxiety in autistic children. This study seeks to address the existing gap in anxiety treatment by examining the feasibility and preliminary efficacy of a novel, telehealth CBT intervention, DINO Strategies for Anxiety and intolerance of Uncertainty Reduction (DINOSAUR), which targets both anxiety and IU in young autistic children.

DETAILED DESCRIPTION:
The purpose of this study is to examine the feasibility and preliminary efficacy of a new treatment that targets both anxiety and IU, i.e., DINOSAUR, in young autistic children with varying cognitive and language levels. To accomplish this goal, we will investigate if DINOSAUR is a feasible intervention for families of young autistic children. We will also investigate if DINOSAUR is superior to an active control condition in reducing anxiety and IU. A third, exploratory goal is to understand how children's language and cognitive level affect their response to anxiety treatment. Seventy children, 4-6 years of age with autism and clinically significant anxiety, and their parents will be randomly assigned to receive either DINOSAUR or the active control (35 in each group) over 14 weeks via telehealth. Within each condition, children will be stratified based on cognitive level. Anxiety and IU will be assessed following treatment and at 4-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 4 years 0 months to 6 years 11 months
* DSM-5 ASD diagnosis based on clinical impressions and results of the Autism Diagnostic Observation Schedule-2 (ADOS-2)
* CBCL Anxiety Problems T-score > 65
* SB-5 ABIQ > 60
* Receptive and expressive language age equivalent > 36 months based on Test of Early Language Development, Fourth Edition (TELD-4)
* Parent (or other caregiver) available and willing to attend 14-week intervention
* Absence of identifiable neurological (e.g., epilepsy), genetic (e.g., Down syndrome, fragile X, tuberous sclerosis, neurofibromatosis) or severe sensory-motor (e.g., severe vision impairment) conditions
* Able to walk independently (a requirement for ADOS-2)

Exclusion Criteria:

* Primary language other than English
* Child is in foster care
* Child displays severe behavior challenges that prevent participation in treatment groups (i.e., severe tantrums, aggression, or self-injury)
* Participating parent experiencing active symptoms of substance abuse or severe mental illness (i.e., schizophrenia, bipolar disorder)

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Change in child anxiety diagnostic status on Anxiety Disorders Interview Schedule, Autism Spectrum Disorder Addendum (ADIS-ASA) | Before and after 14-week treatment (baseline to post-treatment)
  The Anxiety Disorders Interview Schedule (ADIS) is a semi-structured parent interview assessing the severity of anxiety disorders and its presentation in individuals with autism.

SECONDARY OUTCOMES:
Change in anxiety severity on Child Behavior Checklist | Before and after 14-week treatment (baseline to post-treatment) and at 4 month follow-up
  An established 99-item parent and teacher report of broad psychopathology; T scores range from 20 to 100; Syndrome scales: T-scores over 65 indicate clinically significant symptoms.
Change in child's intolerance of uncertainty on Response to Uncertainty and Low Environmental Stability Scale | Before and after 14-week treatment (baseline to post-treatment) and at 4 month follow-up
  Parent and teacher report scale measuring response to uncertainty and low environmental structure; scores range from 1 to 5; higher scores indicate higher intolerance of uncertainty.
Change on parental accommodating behaviors on Family Accommodation Scale following 14-week active control and 14-week intervention. | Before and after 14-week treatment (baseline to post-treatment) and at 4 month follow-up
  Assesses parental accommodating behaviors; scores range from 0 to 36; higher scores indicate higher parental accommodation.

CONTACTS AND LOCATIONS:
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Keefer A, Vasa RA. DINOSAUR: an integrated cognitive-behavioral treatment for anxiety in young children with ASD. J Neurodev Disord. 2021 Oct 11;13(1):46. doi: 10.1186/s11689-021-09396-9. PMID 34635048
- [Result] Vasa RA, Kerns CM, Singh V, McDonald R, Jang YS, Keefer A. Anxiety in autistic preschool children: Phenomenology and a network analysis of correlates. Autism Res. 2023 Aug;16(8):1561-1572. doi: 10.1002/aur.2968. Epub 2023 Jun 23. PMID 37350221